CLINICAL TRIAL: NCT06286358
Title: Impact of Aortic Valve Disease and Thoracic Aortic Aneurysm on Kinocardiographic Signals
Brief Title: Aortopathy Relationship to Imagery and Kinocardiography Features (ARTIK)
Acronym: ARTIK
Status: Recruiting | Type: Observational
Sponsor: Université Libre de Bruxelles (Other)
Collaborators: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Elza Abdessater, Medical doctor at Erasme University Hospital, Erasme University Hospital
Other Study IDs: P2023/346 / CCB : B40620230001
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-03

CONDITIONS: Aortic Valve Disease; Aortic Aneurysm
Keywords: Aortic stenosis; Aortic regurgitation; Thoracic aortic aneurysm; Kinocardiography
MeSH Terms: conditions — Aortic Valve Disease; Aortic Aneurysm; Aortic Valve Stenosis; Aortic Valve Insufficiency; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Interventional treatment: Patients with severe aortic valve disease or thoracic aortic aneurysm in whom interventional treatment has been previously decided by the Heart Team (i.e. the multidisciplinary team of cardiologists and cardiac surgeons treating the patient, independently of the research team) Patients with different severities of AVD or TAA, and healthy subjects. The KCG measurements and video recordings are consecutive to an echocardiography or cardiac MRI, and will be carried out in Erasme hospital.
  Interventions: Diagnostic Test: Kinocardiography
- Aortic valve disease of different severities: Patients with aortic stenosis and/or aortic regurgitation and/or bicuspidy of different severities. The KCG measurements consecutive to the echocardiography and/or cardiac MRI will be carried out during their clinical management in Erasme hospital.
  Interventions: Diagnostic Test: Kinocardiography
- Control: Subjects matched to the two other groups according to their age, gender, body surface area and left ventricular ejection fraction (LVEF), without AVD or TAA. The KCG measurements will be made immediately after the echocardiography and/or MRI in Erasme hospital.
  Interventions: Diagnostic Test: Kinocardiography

INTERVENTIONS:
Diagnostic Test: Kinocardiography — Technology Measuring Cardiac Mechanical Activity Via Accelerometers and Gyroscopes

SUMMARY:
Kinocardiography (KCG) is a portable measurement technique developed to estimate cardiac mechanical performance by studying the vibrations produced by myocardial contraction during each heartbeat and transmitted to the body surface.

The goal of this observational study is to learn about kinocardiography in patients with aortic valve disease (AVD) or thoracic aortic aneurysm (TAA). The investigators believe that this technology will enable to diagnose aortic valve disease and aortic aneurysm.

In patients with AVD of different severities or TAA, the investigators will collect informations from echocardiography and/or cardiac magnetic resonance imaging, KCG recordings, phonocardiography (PCG) recordings, and video recordings. Researchers will also compare subjects without any AVD nor TAA to better understand these effects on KCG, PCG and video signal.

DETAILED DESCRIPTION:
Aortic valve disease (AVD) is a common but under-diagnosed disease which can cause various cardiovascular complications. AVD, including aortic stenosis and aortic regurgitation, can be associated with dilatation of the ascending thoracic aorta as a result of hemodynamic mechanisms and genetic predisposition. In the assessment of an AVD, it is important to consider if it is associated with a thoracic aortic aneurysm (TAA), and vice versa.

The prevalence of TAA in the general population is difficult to assess because most patients are asymptomatic, and their lethal complications (rupture and dissections) are often misdiagnosed as myocardial infarctions. The insidious evolution of aortic pathology motivates physicians to make the diagnosis as early as possible before the appearance of irreversible lesions causing significant morbidity and mortality. Traditional semiology can be useful for AVD screening (auscultation of a murmur, or observation of some visible semiological signs). However, it relies on the proficiency of care providers and may not allow a timely diagnosis of less severe forms of the disease. Moreover, imaging techniques used in current clinical practice are not appropriate for the organization of large-scale screening in asymptomatic patients. In addition, none of these techniques are accessible for the people living far away from a healthcare institution.

Kinocardiography (KCG) is a portable measurement technique developed to estimate cardiac mechanical performance by studying the vibrations produced by myocardial contraction during each heartbeat and transmitted to the body surface. Signals are recorded thanks to a sensor placed on the sternum, another sensor placed on the lower back and electrocardiogram electrodes.

Smartphones are equipped with accelerometers and gyroscope, and may allow anyone to measure their own cardiac mechanical function similarly to KCG.

Phonocardiography (PCG) enables the detailed recording and analysis of heart sounds produced by the blood flow during the opening and closing of heart valves thanks to a microphone. It allows the extraction of heart sound information that reveals valvular diseases, such as the timing of heart valve closure, the frequency content of heart sounds, and the presence of diastolic or systolic murmurs.

Video image processing by Remote photoplethysmography (RPPG) or by Eulerian video magnification (EVM) allow the analysis of color changes and movements, invisible to the naked eye.

The primary objective of this prospective observational study is to better understand and assess KCG signals modifications due to aortic valve disease (AVD) and/or thoracic aortic aneurysm (TAA). It will be possible thanks to imaging techniques such as 4D flow MRI, and thanks to a comparison with PCG. The secondary objective of our study is to evaluate if a smartphone can be used for the diagnostic and characterization of AVD, using KCG, PCG or video image processing.

The possible participants will be identified, according to inclusion/exclusion criteria. Informed consent will be given to the patients. Immediately after the echocardiography and/or the cardiac MRI, the investigators will record KCG and PCG data, and then perform similar measurements using a smartphone placed on the torso. These measurements are followed by two short video recordings of 30 seconds, simultaneously to a KCG recording. For patients undergoing aortic valve replacement or thoracic aortic aneurysm surgery, the investigators will also perform the KCG measurements post-operatively, immediately after de post-operative cardiac MRI and/or echocardiography.

ELIGIBILITY:
Inclusion Criteria

* "Interventional treatment" group

  * Adults (>18 y)
  * Interventional treatment indication for severe AVD and/or severe TAA, as decided by the Heart Team
* "Aortic valve disease of different severities" group

  * Adults (>18y)
  * Aortic stenosis and/or aortic regurgitation and/or bicuspidy of different severities confirmed by echocardiography and/or cardiac MRI
* "Control" group : - Adults (>18 y) appariated with the participants of other groups according to their age, sex, body surface area and LVEF

Exclusion Criteria:

* Any severe rhythm disorder such as frequent ventricular extrasystoles, atrial tachyarrhythmias
* Subject's disabilty to give consent
* Subjects suffering from aortic valve disease or thoracic aortic aneurysm will be excluded from the "control" group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both inpatients and outpatients may be included in "interventional treatment" group and "aortic valve disease of different severities" group.
  "Control" group may include inpatients, outpatients and healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Understand and assess the complex mechanisms underlying the modifications of KCG signals in patients with AVD and/or TAA | 12 months
  Correlation between KCG parameters and imaging parameters (echocardiography, 4D flow MRI)

SECONDARY OUTCOMES:
Comparing KCG to clinical assessment | 18 months
  Correlation between KCG parameters, phonocardiography, semiological signs and video signals
Asses the clinical application of KCG to diagnose AVD and TAA | 18 months
  With a dedicated device and with a smartphone

CONTACTS AND LOCATIONS:
Locations (1):
- Erasme hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No